CLINICAL TRIAL: NCT04033848
Title: Arthroscopically Assisted Treatment of Complex Ankle Fractures - Intraarticular Findings and Prospective PROM Follow-Up
Brief Title: AORIF Complex Ankle Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sebastian. F. Baumbach, Principle Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: AZ 117-15
Record Dates: First submitted 2019-07-19; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Ankle Fractures
Keywords: Arthroscopy; Ankle Fracture; Patient rated outcome
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Arthroscopic assisted ankle fracture treatment — Any complex ankle fracture, as discriped above, will be treated arthroscopically and will be prospectively followed-up using well validated PROMs

SUMMARY:
The aim of this study is to evaluate the intraarticular lesions, to identify fractures specifically at risk for these, and to assess the results following arthroscopically assisted open reduction and internal fixation of complex ankle fractures prospectively.

DETAILED DESCRIPTION:
Starting 05/01/13 patients with complex ankle fractures, older than 17 years, who sustained the injury less than 14 days before surgery and giving informed consent are consecutively enrolled. A complex fracture is defined as either an isolated malleolar fracture in combination with ligamentous instability, or a bi- or trimalleolar fracture. An unstable ligamentous injury is defined as either a disruption of the deltoid ligament leading to increased medial talar tilt, or an unstable syndesmotic injury assessed by the external rotation test both after osteosynthesis of all fractures. Exclusion criteria are isolated unimalleolar fractures, pilon fractures, open fractures, multiple injuries, mental illness, incompliance or pregnancy.

Data assessed are:

* Demographics
* Medical history
* Classification (AO, Haraguchi, ICRS, location and size defect)
* Surgery details
* Complications
* PROMs (FAAM, AOFAS, OMAS, FAOS, TAS, SF-12, EQ-5d, MoxFQ)

ELIGIBILITY:
Inclusion Criteria:

* Unimalleolar fracture + ligamentous injury
* Bi- or trimalleolar fracture ± ligamentous injury
* > 17 years
* Date of injury less than 15 days
* Written informed consent

Exclusion Criteria:

* Isolated unimalleolar fracture
* Pilon fracture
* Open fracture
* Mental illness, incompliance, pregnancy
* Multiple injuries

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient are being recruted from the investigator's ER or foot and ankle outpatient deparment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
OMAS | Through study completion, an average of 1 year
  Olerud and Molander Ankle Score; Validated PROM; Range 0-100

SECONDARY OUTCOMES:
ICRS: Clinical Cartilage Injury Evaluation System | IntraOP
  Intraarticular cartilage lesions and treatment
FAAM | Through study completion, an average of 1 year
  Foot and Ankle Ability Measure, Validated PROM; Range 0-100
AOFAS | Through study completion, an average of 1 year
  American Orthopaedic Foot and Ankle Society, Validated PROM; Range 0-100
FAOS | Through study completion, an average of 1 year
  Foot and Ankle Outcome Score, Validated PROM; Range 0-100
TAS | Through study completion, an average of 1 year
  Tegener Activity Scale, Validated PROM; Range 0-10
SF-12 | Through study completion, an average of 1 year
  Quality of life score, Validated PROM; Range 0-100
EQ-5d | Through study completion, an average of 1 year
  Quality of life score, Validated PROM; Range 0-100
MoxFQ | Through study completion, an average of 1 year
  The Manchester-Oxford Foot Questionnaire, Validated PROM; Range 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Böcker, MD, Study Chair — LMU Munich
Locations (1):
- Department of Trauma Surgery, Medical University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on reasonable demand / colaboration